CLINICAL TRIAL: NCT03289988
Title: Novel Blood-based Colorectal Cancer Screening Method Using Natural Killer Cell Activity and Gene Panel Expression
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2017-0148
Record Dates: First submitted 2017-09-18; First posted 2017-09-21 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Colorectal Adenoma; Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood sampling for genetic analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Normal group: Normal group(control group): patients with negative colonoscopy findings (n= 238).
  Interventions: Other: blood sampling
- Low risk adenoma group: Low risk adenoma group: patients having at least one low risk adenoma (n=250).
  Interventions: Other: blood sampling
- High-risk adenoma group: High-risk adenoma group: patients having at least one of following criteria (more than 1 cm in size, villous or tubulovillous histologic type, high-grade dysplasia findings) (n=316).
  Interventions: Other: blood sampling
- Colon cancer: Colon cancer: histologically confirmed colon cancer patients (n=160).
  Interventions: Other: blood sampling

INTERVENTIONS:
Other: blood sampling — NK activity and gene panel expression analysis based on blood test (5cc blood sampling)

SUMMARY:
Natural killer cells (NK cells) are cytotoxic lymphocytes that play an important role in the innate immune system. In particular, it plays a very important defense function against host cells or cancer cells infected with a specific virus. Recent studies have shown that the activity of NK cells is decreased in patients with various carcinomas compared with normal controls, suggesting that the measurement of activity of NK cells in the blood may be helpful in the early diagnosis of cancer. In a recent study analyzing NK cell activity in 762 patients undergoing colonoscopy, NK cell activity showed performance in diagnosing advanced colorectal adenoma and colorectal cancer with sensitivities 42.2% and 85.7%, and specificity 58.3% and 59.5%, respectively. This finding suggests that NK cell activity may be useful as a screening method for colorectal neoplasms. However, as a single test, this diagnostic power is relatively low. On the other hands, another blood-based colorectal cancer screening test that using 29 gene panels algorithm has recently been reported. According to this study, 29 gene panel algorithms (Colox®) showed performance in diagnosing advanced colorectal adenoma and colorectal cancer with sensitivity of 55.4% and 79.5% and specificity of both 90.0%, respectively. for diagnosis of advanced adenoma and colorectal cancer, respectively. Although the Colox® test seems to be useful for the colorectal cancer screening using blood test, this diagnostic power is relatively low. In order to overcome low diagnostic performance of aforementioned tests (NK activity and Colox®) as a single use, combination of individual biomarkers can be a promising alternative. In this regards, the aim of this study was to evaluate the diagnostic value for predicting advanced colorectal neoplasms by combining Colox® and NK cell activity indicators.

ELIGIBILITY:
Inclusion Criteria:

* Adults population over 40 years of age
* Patients who understood this study process and agreed to participation of this study
* Colon cancer patients who have been confirmed as colorectal cancer by endoscopic biopsy within 1 month
* Colon cancer patients who received no anticancer treatment such as surgery, chemotherapy, radiation therapy after cancer diagnosis.
* Colorectal adenoma and normal control group: Patients undergoing colonoscopy for diagnostic purposes or colorectal cancer screening.

Exclusion Criteria:

* Patients who did not agree to participate in the study and did not write their informed consent
* Vulnerable subjects with mental retardation or severe psychiatric illness.
* Patients who are not appropriate enrollment of this study by researchers judgement.
* Patients who have had an immunosuppressive drug within 6 months.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Normal group: patients with negative colonoscopy findings (n= 238).
  2. Low risk adenoma group: patients having at least one low risk adenoma (n=250).
  3. High-risk adenoma group: patients having at least one of following criteria (more thatn 1 cm in size, villous or tubulovillous histologic type, high-grade dysplasia findings) (n=316).
  4. Colon cancer: histologically confirmed colon cancer patients (n=160).
Sampling Method: Probability Sample
Enrollment: 964 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Power for prediction of advanced colorectal neoplasms | 2 months
  Diagnostic Power for prediction of advanced colorectal neoplasms using combination of conventional Colox® and NK Cell Activity Indicators.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Internal Medicine, Yonsei University College of Medicine, Seoul, South Korea